CLINICAL TRIAL: NCT05029011
Title: Low-cost Sensor System for COVID-19 Patient Monitoring: Validation of BRAEBON Vital Signs Monitor (VTS)
Status: Completed | Type: Observational
Sponsor: Helen S. Driver, PhD (Other)
Collaborators: Braebon Medical Corporation (Unknown); National Research Council, Canada (Unknown)
Responsible Party: Sponsor-Investigator, Helen S. Driver, PhD, Dr. Helen S. Driver, Assistant Professor, Division of Respirology and Sleep Medicine, Dept. Medicine, Queen's University, Queen's University
Organization: Queen's University (Other)
Other Study IDs: DMED-2496-21
Record Dates: First submitted 2021-08-16; First posted 2021-08-31 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients of the Sleep Disorders Laboratory: Monitoring vital signs
  Interventions: Device: BRAEBON VTS

INTERVENTIONS:
Device: BRAEBON VTS — The BRAEBON VTS is a portable device that continuously monitors vital signs. Participants in the study will wear the BRAEBON VTS for 24 hours.

SUMMARY:
The BRAEBON VTS is a low-cost, portable device that is being developed to take continuous and real-time vital sign measurements of COVID-19 patients, both in the hospital and home setting. This study is being undertaken to test the BRAEBON VTS and validate against industry standards.

DETAILED DESCRIPTION:
In response to the COVID-19 pandemic, the BRAEBON Vital Signs Monitor (VTS) has been developed with funding from the National Research Council of Canada Industrial Research Assistance Program through the federal government's Innovative Solutions Canada (ISC) program. The VTS will measure peripheral capillary oxygen saturation (SpO2) and pulse via photoplethysmography (PPG), temperature, blood pressure (BP), heart and respiration rates, electrocardiogram (ECG), head position and movement over a continuous period. This monitor can be used remotely, and importantly will be low-cost so it can be accessed widely. Data from the VTS is transmitted wirelessly to a portable basestation which is a smartphone or tablet device via a customized application. This study will test the VTS both within the clinical environment and in the remote home environment to see how well it monitors patients effected by COVID-19 needing care, as well as satisfying an unmet need for remote monitoring across the healthcare system.

This study will compare the newly developed VTS with an industry gold standard of polysomnography (PSG) in the sleep laboratory, or in the home with the MediByte Jr (home sleep apnea test).

Approximately 150 patients will be recruited to the study across two different settings which includes a hospital setting and a remote setting, within the home environment.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a sleep evaluation using polysomnography
* People referred to the sleep clinic
* Persons over the age of 18

Exclusion Criteria:

* Unable and/or unwilling to consent
* No access to home WIFI (applicable to participants local to Kingston undertaking the study in the home setting)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of who under the care of the sleep disorders lab
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Oximetry - overnight comparison between the VTS and gold-standard PSG | Up to 24 hours (Overnight - between lights-off and lights-on as for standard overnight sleep recordings).
  Time spent with oxygen saturation >=90%, time spent with oxygen saturation <= 88%, number of desaturations of >3%
Cardiac Rate (heart rate/pulse) | Up to 24 hours (Overnight - between lights-off and lights-on as for standard overnight sleep recordings).
  beats per minute
Blood Pressure (BP) | evening and morning, in a 24 hour period
  mmHg
Temperature (forehead) | evening and morning, in a 24 hour period
  degrees celcius
Body position (PSG and MediByte Jr) and head position (VTS) | Up to 24 hours (Overnight - between lights-off and lights-on as for standard overnight sleep recordings).
  minutes spent supine, lateral and prone
Respiratory rate | Up to 24 hours (Overnight - between lights-off and lights-on as for standard overnight sleep recordings).
  breaths per minute
Identification of artifact | Up to 24 hours (Overnight - between lights-off and lights-on as for standard overnight sleep recordings).
  e.g. movement

SECONDARY OUTCOMES:
Develop guidelines for the VTS | Within 6 months
  After assessing the usability of the VTS in the sleep laboratory and remote use in the home.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Driver, Phd, Principal Investigator — Queen's University and Kingston Health Sciences Centre
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No